CLINICAL TRIAL: NCT02658422
Title: An Open-label Balanced, Randomised, Single Dose, Two-way Crossover Study to Determine the Bioequivalence of GW483100 10 mg Tablets (Containing Montelukast Sodium Equivalent to 10 mg of Montelukast) Relative to Reference Montelukast Sodium 10 mg Tablets (Containing Montelukast Sodium Equivalent to 10 mg of Montelukast) in Healthy Male and Female Volunteers Under Fasting Conditions
Brief Title: Bioequivalence of GW483100 10 Milligram (mg) Tablets in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201681
Record Dates: First submitted 2015-07-06; First posted 2016-01-18 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Disorders; Asthma and Rhinitis
MeSH Terms: conditions — Respiration Disorders; Asthma; Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A-B (Test Montelukast then Reference Montelukast) (Experimental): Subjects will receive Treatment A- Test montelukast sodium 10 mg tablets (GW483100) in Treatment Period 1 and then Treatment B - Reference montelukast sodium 10 mg tablets (innovator product) in Treatment Period 2.
  Interventions: Drug: Test Montelukast; Drug: Reference Montelukast
- Sequence B-A (Reference Montelukast then Test Montelukast) (Experimental): Subjects will receive Treatment B- Reference montelukast sodium 10 mg tablets (innovator product) in Treatment Period 1 and then Treatment A Test montelukast sodium 10 mg tablets (GW483100) in Treatment Period 2.
  Interventions: Drug: Test Montelukast; Drug: Reference Montelukast

INTERVENTIONS:
Drug: Test Montelukast — Test Montelukast (GW483100) is available as round, biconvex, pink 10 mg film-coated tablet (containing montelukast sodium equivalent to 10 mg of montelukast) and is administered as a single dose with 240 mL of water.
Drug: Reference Montelukast — Reference Montelukast (innovator product) is available as pale beige, rounded square shaped,10 mg film-coated tablet (containing montelukast sodium equivalent to 10 mg of montelukast) and is administered as a single dose with 240 mL of water. Singular is the innovator product used for this study, which is a trade name owned by Merck Sharp and Dohme Corporation.

SUMMARY:
This study is conducted to determine whether the test product (GW483100 10 mg containing montelukast sodium equivalent to 10 mg of montelukast) is bioequivalent to the reference montelukast sodium 10 mg tablets (innovator product) in healthy adult volunteers under fasting conditions. This is an open-label, balanced, randomized, single dose, two-way crossover study, enrolling 32 healthy human subjects to ensure at least 28 subjects complete the study. Each subject enrolled will participate in two treatment periods separated by a washout period of at least 7 days and no more than 14 days between dosing occasions. Total duration in the study for each subject will be approximately 7 weeks from screening to the subject's last visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy, non smoker, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 19 - 24.9 kg/square meter (m^2) (inclusive)
* Healthy male or female subjects: MALES: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 24 hours after the last dose of study medication. a.) Vasectomy with documentation of azoospermia. b.) Male condom plus partner use of one of the contraceptive following options: contraceptive subdermal implant; intrauterine device or intrauterine system; oral contraceptive, either combined or progestogen alone; injectable progestogen; contraceptive vaginal ring; and percutaneous contraceptive patches. FEMALES: Eligible to participate, if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: a.) Non-reproductive potential defined as: Pre-menopausal females with one of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, Documented Bilateral Oophorectomy Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. b.) Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until 24 hours after the last dose of study medication and completion of the follow-up visit.
* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT (QTc) > 450 millisecond (msec) NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read; The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial; For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).
* No concomitant medications should be taken by the subject while participating in the study.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 90 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* Any symptoms with a systolic BP <95 millimeter of mercury (mmHg).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2015-09-21 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time from time zero to infinity (AUC(0 ∞)) for montelukast in relevant treatments | Samples will be collected at Pre-dose, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post-dose in each treatment period
  Blood samples will be withdrawn on Day 1 and Day 2, and concentrations of montelukast will be determined in plasma samples. Plasma montelukast concentration-time will be analyzed by non-compartmental method and the PK parameters will be derived.
AUC from time zero to last time point with measurable concentration (AUC(0-t)) for montelukast in relevant treatments | Samples will be collected at Pre-dose, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post-dose in each treatment period
  Blood samples will be withdrawn on Day 1 and Day 2, and concentrations of montelukast will be determined in plasma samples. Plasma montelukast concentration-time will be analyzed by non-compartmental method and the PK parameters will be derived.
Maximum observed concentration (Cmax) for montelukast in relevant treatments | Samples will be collected at Pre-dose, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post-dose in each treatment period
  Blood samples will be withdrawn on Day 1 and Day 2, and concentrations of montelukast will be determined in plasma samples. Plasma montelukast concentration-time will be analyzed by non-compartmental method and the PK parameters will be derived.

SECONDARY OUTCOMES:
Time of occurrence of Cmax (tmax) for montelukast in relevant treatments | Samples will be collected at Pre-dose, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post-dose in each treatment period.
  Blood samples will be withdrawn on Day 1 and Day 2, and concentrations of montelukast will be determined in plasma samples. Plasma montelukast concentration-time will be analyzed by non-compartmental method and the PK parameters will be derived.
Percentage of AUC(0-∞) obtained by extrapolation (%AUCex) for montelukast in relevant treatments | Samples will be collected at Pre-dose, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post-dose in each treatment period.
  Blood samples will be withdrawn on Day 1 and Day 2, and concentrations of montelukast will be determined in plasma samples. Plasma montelukast concentration-time will be analyzed by non-compartmental method and the PK parameters will be derived.
Terminal phase half-life (t½) for montelukast in relevant treatments | Samples will be collected at Pre-dose, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post-dose in each treatment period.
  Blood samples will be withdrawn on Day 1 and Day 2, and concentrations of montelukast will be determined in plasma samples. Plasma montelukast concentration-time will be analyzed by non-compartmental method and the PK parameters will be derived.
Blood pressure (BP) as a measure of safety and tolerability | 3 days in each treatment period (assessed up to 3 weeks)
  Systolic and diastolic BP will be measured in supine position after 5 minutes rest.
Pulse rate measurements as a measure of safety and tolerability | 3 days in each treatment period (assessed up to 3 weeks)
  Pulse rate measurements will be measured in supine position after 5 minutes rest.
Number of participants with adverse events (AEs) | Up to 7 weeks
  AEs will be collected from the start of study treatment until the subject's last visit.
Composite of hematology parameters as a measure of safety | 1 day in Treatment Period 1 and 2 days in Treatment Period 2 (assessed up to 3 weeks)
Composite of clinical chemistry parameters as a measure of safety | 1 day in Treatment Period 1 and 2 days in Treatment Period 2 (assessed up to 3 weeks)
Composite of urinalysis parameters as a measure of safety | 1 day in Treatment Period 1 and 2 days in Treatment Period 2 (assessed up to 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Telangana, India

REFERENCES:
- See also: Results for study 201681 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201681?search=study&b'search_terms=201681'#rs